CLINICAL TRIAL: NCT03210974
Title: Retrospective Observational Study About the Evolution of Patients With Breast Cancer in Hospitals From the GEICAM Group (2002 - 2005). ALAMO IV
Brief Title: Retrospective Observational Study About Evolution of Patients With Breast Cancer in Hospitals From GEICAM Group
Acronym: ALAMO-IV
Status: Completed | Type: Observational
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Other Study IDs: ÁLAMO IV
Record Dates: First submitted 2017-06-19; First posted 2017-07-07 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Invasive Breast Cancer Between 2002 and 2005

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a non-interventional (NIS), multicenter, retrospective cohort study, which will obtain data from patients diagnosed with invasive breast cancer between 2002 and 2005 in the medical oncology departments of hospitals that are members of GEICAM (using information obtained from patient medical histories).

DETAILED DESCRIPTION:
There is no specific treatment regimen for this study. This is an observational retrospective study in which the clinical decisions concerning the optimal strategy in the treatment of the disease for each patient have been taken independently and prior to the physician's decision to include patient data in this registry, in keeping with the drug information, local treatment guidelines and/or standard clinical practice.

The study target population are all patients (men and women) who have been newly diagnosed with invasive breast cancer between January 1, 2002 and December 31, 2005 and treated in the medical oncology departments of participating sites, ensuring an approximate follow-up of 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose first primary breast invasive tumor diagnosis occurred between January 1, 2002 and December 31, 2005 and who have received treatment in the medical oncology departments of participating sites.
* Patients who were diagnosed at the participating site; otherwise the site where the initial diagnosis was made should be contacted with in order to confirm that the patient has not already been enrolled in the study or pending inclusion. The objective is to avoid duplicate records for displaced patients.

Exclusion Criteria:

* Patients with a single diagnosis of in situ carcinoma (without infiltrating component).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study target population are all patients (men and women) who have been newly diagnosed with invasive breast cancer between January 1, 2002 and December 31, 2005 and treated in the medical oncology departments of participating sites, ensuring an approximate follow-up of 10 years.
Sampling Method: Non-Probability Sample
Enrollment: 13135 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Study demographic | 30 months
  Number of participants with the demographic characteristics: Age, sex, race of new cases of breast cancer diagnosed from 2002 to 2005 in Spanish hospitals.
Study clinical and anatomic-pathological | 30 months
  In the 12.000 patients included to study the clinical and anatomic-pathological characteristics: primary tumor, regional nodes, metastasis status (TNM), date of initial diagnosis of Breast Cancer (BC), biomarkers of new cases of breast cancer diagnosed from 2002 to 2005 in Spanish hospitals

SECONDARY OUTCOMES:
Evolution of Breast Cancer in terms of frequency | 30 months
  In the 12.000 patients included to describe the evolution of breast cancer patients in terms of frequency (time).
Evolution of Breast Cancer in terms of type | 30 months
  In the 12.000 patients included to describe the evolution of breast cancer patients in terms of type of relapse.
Evolution of Breast Cancer in terms of location of relapse | 30 months
  In the 12.000 patients included to describe the evolution of breast cancer patients in terms of location of relapse.
Family history of Breast Cancer | 30 months
  Number of patients with a family history of breast cancer.
Characteristics of family history of Breast Cancer | 30 months
  Characteristics clinical-pathological of patients with a family history of breast cancer.
Differences in Breast Cancer between sex | 30 months
  Differences clinical-pathological between men and women with breast cancer
Quantify the influence of type of surgery conducted on primary tumor | 30 months
  In the 12.000 patients included to quantify the influence of type of surgery conducted on primary tumor
Number of patients with metastatic disease as first diagnosis | 30 months
  In the 12.000 patients included to quantify the influence of timepoint of primary tumor surgery in patients with metastatic disease as first diagnosis
Quantify the prevalence of breast cancer related to pregnancy | 30 months
  In the 12.000 patients included to quantify the prevalence of breast cancer related to pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital Universitario Fundación Alcorcón; Study Director, Study Director — Hospital General Universitario Gregorio Marañón; Study Director, Study Director — Instituto de Salud Carlos III de Madrid
Locations (41):
- Spain (41):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital General Universitario de Elda - Virgen de la Salud, Elda, Alicante
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital General de Granollers, Granollers, Barcelona
  - Hospital de Mataró-Consorci Sanitari del Maresme, Mataró, Barcelona
  - Corporació Sanitaria Parc Taulí, Sabadell, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Onkologikoa, Donostia / San Sebastian, Guipuzcoa
  - Hospital Universitario de Donostia, Donostia / San Sebastian, Gupúzcoa
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Fundación Alrcorcón, Alcorcón, Madrid
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda, Madrid
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Virgen de los Lirios, Alcoy, Valencia
  - Hospital Universitario de Basurto, Bilbao, Vizcaya
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Centro Oncológico de Galicia, A Coruña
  - Complejo Hospitalario de Albacete, Albacete
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Nuestra Señora de Sonsoles, Ávila
  - Hospital del Mar, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital General Virgen de la Luz, Cuenca
  - Hospital Josep Trueta, Girona
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario La Prinesa, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Complejo Hospitalario Universitario de Ourense, Ourense
  - Hospital Universitario Virgen de la Salud, Toledo
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Universitari i Politécnic La Fe, Valencia
  - Hospital Clínico Universitario de Zaragoza Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lopez-Tarruella S, Escudero MJ, Pollan M, Martin M, Jara C, Bermejo B, Guerrero-Zotano A, Garcia-Saenz J, Santaballa A, Alba E, Andres R, Martinez P, Calvo L, Fernandez A, Batista N, Llombart-Cussac A, Anton A, Lahuerta A, de la Haba J, Lopez-Vega JM, Carrasco E. Survival impact of primary tumor resection in de novo metastatic breast cancer patients (GEICAM/El Alamo Registry). Sci Rep. 2019 Dec 27;9(1):20081. doi: 10.1038/s41598-019-55765-9. PMID 31882586
- See also: Spanish Breast Cancer Research Group (GEICAM) is a Spanish Breast Cancer Research Group — http://www.geicam.org